CLINICAL TRIAL: NCT03533036
Title: Feasibility of an Immersive Virtual Reality Intervention for First Trimester D&C: A Pilot Study
Brief Title: Virtual Reality Experience in First Trimester D&C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Aparna Sridhar, MD, MPH, FACOG, Assistant Professor in Obstetrics and Gynecology at David Geffen School of Medicine at UCLA, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB#17-001122
Record Dates: First submitted 2018-03-12; First posted 2018-05-22 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: First Trimester Abortion; Virtual Reality
Keywords: Virtual Reality; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Time series study with 15 controls and 15 experimental group. Investigators plan to enroll 30 patients in order to obtain an effect size for future studies. The mean and standard deviation of anxiety scores for each group will be used to calculate power for future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virtual Reality Intervention (Experimental): VR headsets consist of a Samsung phone dedicated to playing programs designed by the AppliedVR company. The phone is inserted in the front of the headset and can play videos that can be then viewed by the participant while wearing the headset. Participants in the experimental arm will be fitted with VR headsets prior to first trimester abortion and will wear the headset during the procedure. Participants will be able to choose a program of their preference (ex. guided meditation, beautiful scenery). The patient may remove the VR device at any time during the procedure. After the procedure, investigators will carry out a qualitative interview with the participant and ask about the experience of using the VR headset during first trimester abortion. Patients will also complete surveys evaluating procedure-related anxiety. These will be administered before and after the procedure.
  Interventions: Device: applied VR headset
- Control arm (No Intervention): In the control group, participants will not use virtual reality during the procedure. Patients in the control arm will complete surveys evaluating procedure-related anxiety. These will be administered before and after the procedure.

INTERVENTIONS:
Device: applied VR headset — Virtual reality (VR) is a three-dimensional experience created by a headset fitted with a video display. The device, designed to be worn on the face, immerses the viewer in a virtual world and can create a visual distraction from the patient's present situation. We will use a commercially available VR device, comprised of a phone and headset. The phone is inserted into the headset to act as the visual display that can create three dimensional environments. The patient will then choose the virtual reality experience she prefers from the two relaxation programs available. The VR device will be introduced to the participant and fitted to her head prior to the procedure. The device is intended to be worn during the full length of the procedure until the conclusion of the D&C, however the participant may decide to stop wearing the device and choose to end the VR experience at any time.
  Arms: Virtual Reality Intervention

SUMMARY:
Virtual reality (VR) has been used in health care settings to decrease anxiety and pain. This project is a feasibility study to evaluate whether virtual reality can be used in the setting of a first trimester pregnancy termination by D&C and whether the use of virtual reality (VR) headsets can help decrease anxiety for patients during this procedure.

DETAILED DESCRIPTION:
The investigators will assess the practicality and qualitative experience of women using VR during first trimester surgical abortion under local anesthesia. Semi-structured interviews will be conducted to understand the patient's experience of using VR. Surveys evaluating anxiety will be administered to women before and after surgical abortion. Investigators plan to enroll 30 patients in order to obtain an effect size for future studies. A group of control patients will be enrolled; these patients will receive standard care and will be compared to the anxiety scores of the group receiving VR. The mean and standard deviation of anxiety scores for each group will be used to calculate power for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Elective surgical abortion under local anesthesia
* English speaker

Exclusion Criteria:

* No psychiatric history
* No history of motion sickness or vertigo
* No history of seizures or epilepsy
* No recent eye surgery or visual impairment
* No claustrophobia.
* No current nausea or vomiting
* Not on seizure-threshold lowering medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be biologically female, willing to have a first trimester abortion
Enrollment: 30 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles Obstetrics and Gynecology Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757
- [Background] Shourab NJ, Zagami SE, Golmakhani N, Mazlom SR, Nahvi A, Pabarja F, Talebi M, Rizi SM. Virtual reality and anxiety in primiparous women during episiotomy repair. Iran J Nurs Midwifery Res. 2016 Sep-Oct;21(5):521-526. doi: 10.4103/1735-9066.193417. PMID 27904638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants recruited to each group (experimental vs control)
Pre-assignment Details: Patients were assigned to either experimental or control group via convenient sampling.
Groups:
- Virtual Reality Intervention: Participants in the experimental arm were fitted with VR headsets prior to first trimester abortion and could choose to wear the headset during the procedure. Participants chose a program of their preference (ex. guided meditation, beautiful scenery). The patient was able to remove the VR device at any time during the procedure.
- Control Arm: In the control group, participants did not use virtual reality during the procedure.
Period: Overall Study
Arm/Group | Virtual Reality Intervention | Control Arm
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Intervention | Control Arm | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6.9) | 31 (7.8) | 30 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 5 | 5 | 10
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Able to Use VR Device Throughout the Entire Duration of First Trimester Surgical Abortion.
Description: Number of participants able to use VR device throughout the entire duration of first trimester surgical abortion.
Time Frame: 15 minutes
Measure: Number; unit: participants
Arm/Group | Virtual Reality Intervention
Number analyzed (Participants) | 15
participants | 6

2. Secondary Outcome: Change in Procedure Related Anxiety as Assessed by the Visual Analog Scale (VAS).
Description: Mean change in procedure related anxiety score as assessed by the Visual Analog Scale (VAS).
  The Visual Analog Scale is a 11 point scale ranging from 0 to 10. 0 indicates the least amount of discomfort or anxiety whereas 10 represents the most amount of discomfort or anxiety.
  Participants were surveyed on their level of discomfort prior to and after the procedure. The difference of these scores was taken and the average of each group is presented in as a result.
Time Frame: 30 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Intervention | Control Arm
Number analyzed (Participants) | 15 | 15
units on a scale | -3.97 (3.20) | -2.71 (2.89)

ADVERSE EVENTS:
Time Frame: During period of participant enrollment and data collection (45 minutes)
Arm/Group | Virtual Reality Intervention | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT03533036/Prot_SAP_000.pdf